CLINICAL TRIAL: NCT06301256
Title: An Open-label Single Center Study to Evaluate the Efficacy of TIRZEPATIDE for the Treatment of Moderate to Severe Hidradenitis Suppurativa
Brief Title: Evaluate the Efficacy of TIRZEPATIDE for the Treatment of Moderate to Severe HS Hidradenitis Suppurativa
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida Academic Centers Research and Education, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I8F-NS-I002
Record Dates: First submitted 2024-03-01; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — Tirzepatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: TIRZEPATIDE — Tirzepatide injection contains tirzepatide, a once weekly dual receptor, GIP and GLP-1 receptor agonis t. It is a 39-amino-acid modified peptide with a C20 fatty diacid moiety that enables albumin binding and prolongs the half-life. The molecular weight is 4813.53 Da and the empirical formula is C225H348N48O68.

SUMMARY:
The purpose of this study is to determine the clinical efficacy and safety of tirzepatide in subjects with moderate to severe hidradenitis suppurativa. The study will be conducted over 24 weeks on active therapy followed by a eight-week observational follow-up visit. The total length of the study will be 32 weeks .

ELIGIBILITY:
Inclusion Criteria:

Written informed consent provided by the patient. Male or female, age 18 years. BMI of 27 or greater Subject must be in general good health (except for hidradenitis suppurativa) as judged by the investigator, based on medical history, physical examination, clinical laboratories, and urinalysis. NOTE: the definition of good health means a subject that does not have uncontrolled significant co-morbid conditions.

Must have a diagnosis of HS for at least 6 months prior to Baseline/Screening visit Subjects with moderate to severe HS with a PGA score of 3 or more. 3 is defined as having: 0 abscesses, 0 draining fistula, and 5 inflammatory nodules; or 1 abscess or draining fistula and 1 inflammatory nodule; or 2-5 abscesses or draining fistulas and 10 inflammatory nodules. Patients with more than 5 abscesses or 5 draining fistulas, and/or excessive scarring, will be excluded.

HS lesions must be present in at least two distinct anatomic areas, one of which must be at least Hurley Stage II (see definition of terms) Subject must have stable HS for at least 2 months (60 days) prior to Screening/Baseline visit as determined by the investigator through subject interview and review of medical history.

Subject must agree to daily use (and throughout the entirety of the study) of one of the following over-the- counter topical antiseptics on their HS lesions: chlorhexidine gluconate, triclosan, benzoyl peroxide, or dilute bleach in bathwater.

Premenopausal women must have a negative serum pregnancy test on entry in the study.

Women who are post-menopausal will have their FSH checked to confirm their status.

Females of childbearing potential (FCBP)† must have a negative pregnancy test at Screening and Baseline. While on investigational product and for at least 28 days after taking the last dose of investigational product, FCBP who engage in activity in which conception is possible must use one of the approved contraceptive options described below:

Option 1: Any one of the following highly effective methods: hormonal contraception (injection, implant, transdermal patch, vaginal ring); intrauterine device (IUD); tubal ligation; or partner's vasectomy; OR Option 2: Male or female condom (latex condom or nonlatex condom NOT made out of natural [animal] membrane [for example, polyurethane]; PLUS, one additional barrier method: (a) diaphragm with spermicide; (b) cervical cap with spermicide; or (c) contraceptive sponge with spermicide d) oral hormonal contraception.

Use of Tirzepatide may reduce the efficacy of oral hormonal contraceptives due to delayed gastric emptying. This delay is largest after the first dose and diminishes over time. Advise patients using oral hormonal contraceptives to switch to a non-oral contraceptive method, or add a barrier method of contraception for 4 weeks after initiation and for 4 weeks after each dose Escalation with tirzepatide.

Male subjects (including those who have had a vasectomy) who engage in activity in which conception is possible must use barrier contraception (male latex condom or nonlatex condom NOT made from natural [animal] membrane [for example, polyurethane]) while on investigational product and for at least 28 days after the last dose of investigational product.

A female of childbearing potential is a sexually mature female who 1) has not undergone a hysterectomy (the surgical removal of the uterus) or bilateral oophorectomy (the surgical removal of both ovaries) and 2) has not been postmenopausal for at least 24 consecutive months (that is, has had menses at any time during the preceding 24 consecutive months).

The female subject's chosen form of contraception must be effective by the time the female subject is screened into the study (for example, hormonal contraception should be initiated at least 28 days before screening).

The screening/baseline laboratory test results must meet the following criteria (WNL means within normal limits for patients with HS [e.g., may have slightly higher WBC and platelet counts]):

* WBC (white blood cell count): WNL
* ANC (absolute neutrophil count): WNL
* Hemoglobin: >10 mg/dl
* Platelets: WNL
* Serum Creatinine: WNL
* SGOT (AST - aspartate aminotransferase): <3 times upper normal limit
* SGPT (ALT - alanine aminotransferase): <3 times upper normal limit
* Alkaline phosphatase:<3 times upper normal limit
* FSH for postmenopausal women (to confirm menopause has occurred and exclude the need for contraception)

Exclusion Criteria:

Subjects with 20 nodular lesions and/or significant scarring (defined as any linear, indurated area, extended across more than 50% of the circumference of the affected area), more than 5 abscesses, more than 5 fistulas or sinus tracts.

Patient with PGA 0-2 (no disease or minimal disease i.e.: Hurley Stage 1) will be excluded.

Patients with BMI lower than 27 Patients with a personal or family history of MTC or in patients with Multiple Endocrine Neoplasia syndrome type 2 (MEN 2).

Patients with Type 1 Diabetes Mellitus History of pancreatitis Other than hidradenitis suppurativa, any clinically significant (as determined by the investigator) cardiac, endocrinologic, pulmonary, neurologic, psychiatric, hepatic, renal, hematologic, immunologic disease, or other major disease that is currently uncontrolled.

Any condition, including the presence of laboratory abnormalities, which would place the subject at unacceptable risk if he/she were to participate in the study. Prior history of suicide attempt at any time in the subject's lifetime prior to or major psychiatric illness requiring hospitalization within the last 3 years.

Women who are pregnant, nursing, or planning pregnancy within 6 months after the last study drug dose (this includes fathers who plan on fathering a child within 6 months after their last study drug dose.

Known serious hypersensitivity to tirzepatide or any of the excipients in it. Serious hypersensitivity reactions, including anaphylaxis and angioedema, have been reported with tirzepatide.

Active substance abuse or a history of substance abuse within 6 months prior to Screening Malignancy or history of malignancy, except for treated [i.e., cured] basal cell or squamous cell in situ skin carcinomas; treated [i.e., cured] cervical intraepithelial neoplasia (CIN) or carcinoma in situ of cervix with no evidence of recurrence within the previous 5 years.

Active substance abuse or a history of substance abuse within 6 months prior to screening Patient with diagnosis or suspected Crohn's disease or ulcerative colitis. Patient who is on a stable dose of analgesics, will be allowed to remain on them. No new opiates will be permitted during the trial.

Use of any investigational drug within 5 weeks prior to screening, or 5 pharmacokinetic/pharmacodynamic half-lives, if known (whichever is longer).

Known allergy to tirzepatide, semaglutide, exenatide, liraglutide or other incretins (GLP1 receptor agonists) Have a known history of serious infections (i.e, hepatitis, pneumonia or pyelonephritis) in the previous 3 months Have a history of lymphoproliferative disease, including lymphoma or signs suggestive of possible lymphoproliferative disease such as lymphadenopathy of unusual size or location (eg, nodes in the posterior triangle of the neck, infraclavicular, epitrochlear, or periaortic area), or splenomegaly Have current signs or symptoms of severe, progressive, or uncontrolled renal, hepatic, hematologic, gastrointestinal, endocrine, pulmonary, cardiac, neurologic, or cerebral disease.

Are unable or unwilling to undergo multiple venipunctures because of poor tolerability or lack of easy access.

Patient with significant scarring, fistulas, or sinus tract involvement will be excluded. Only subjects with inflammatory abscesses and nodules will be allowed to enter the study.

Infection(s) requiring treatment with intravenous (IV) anti-infectives (antibiotics, antivirals, antifungals) within 30 days prior to Baseline or oral anti-infectives (antibiotics, antivirals, antifungals) within 14 days prior to Baseline.

Any other active skin disease or condition (e.g., bacterial, fungal or viral infection) that may interfere with assessment of HS; History of invasive infection (e.g., listeriosis, histoplasmosis), human immunodeficiency virus (HIV); Subject has an active systemic viral infection or any active viral infection that based on the investigator's clinical assessment make the subject an unsuitable candidate for the study; Hepatitis B: HBsAg positive (+) or detected sensitivity on the HBV-DNA PCR qualitative test for HBc Ab/HBsAb positive subjects; Or Hepatitis C Have evidence of active or Latent TB Pregnant (or considering becoming pregnant) or lactating females. Subjects currently undergoing any of the following treatments for HS will require a 4 week wash- out period: minocycline; tetracycline; clindamycin; rifampin and steroids. Patients treated with any biologic therapy including adalimumab, will require a washout period of 5 half lives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03-11 (Estimated); Primary Completion 2025-03-11 (Estimated); Study Completion 2025-03-11 (Estimated)

PRIMARY OUTCOMES:
Hidradenitis Suppurativa Clinical Response (HiSCR) 50% | 24 Weeks
  The proportion of subjects achieving Hidradenitis Suppurativa Clinical Response (HiSCR) at week 24, defined as a 50% reduction in the total number of inflammatory nodule count, as long as the number of fistulae and abscesses don't increase.

IPD SHARING:
Plan to Share IPD: No